CLINICAL TRIAL: NCT01411280
Title: Ameliorating Attention Problems in Children With SCD
Brief Title: Ameliorating Attention Problems in Children With Sickle Cell Disease (SCD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R21HD049244-01 (NIH)
Record Dates: First submitted 2006-07-20; First posted 2011-08-08 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2011-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Laboratory trial (Placebo Comparator): Compare methylphenidate to placebo in an acute laboratory trial
  Interventions: Drug: methylphenidate
- Home/School trial (Experimental): Low dose and moderate dose methylphenidate are compared to placebo in a home and school trial
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Drug: methylphenidate — Ritalin 10mg, Ritalin 20mg
  Other Names: Ritalin

SUMMARY:
The purpose of this study is to assess whether methylphenidate is effective in enhancing the cognitive performance of children with the HbSS or HbSC genotype of SCD who have sustained neurological complications on laboratory-based measures of sustained attention, reaction time, and executive functions, and indirectly, verbal short-term and long-term memory.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a group of autosomal recessive disorders, affecting an estimated 1 in 400 African American newborns annually. The pathophysiology of this group of disorders involves the production of abnormal hemoglobin (HbS), which causes red blood cells to assume a rigid, sickled shape upon release of oxygen, thereby reducing their viability in circulation. Consequently, chronic anemia and system-wide ischemia result in acute painful episodes, organ system failure, and neurological complications. Among the most debilitating effects of SCD are neurological complications. Despite the mounting evidence for structural and functional involvement of the frontal systems in pediatric SCD, there have been no clinical trials designed to manage the cognitive and behavioral sequelae associated with pediatric SCD.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent can be obtained from parent or care-giver and Assent can be obtained from the child
* Children with sickle cell disease (HbSS or HbSC)
* Age range from 6 to 16 years inclusive
* English is the child's primary language
* T-score greater than or equal to 63 on either the Conners' Parent Rating Scale - Revised or the Conners' Teacher Rating

Exclusion Criteria:

* History of glaucoma for which methylphenidate is contraindicated
* Child or immediate family member has a history of a tic disorder or Tourette's syndrome
* Child is currently receiving antidepressant, anxiolytic, antipsychotic, or stimulant drug therapy
* Family history of substance abuse disorder due to potential for abuse of stimulants by caregivers or other family members
* Recent history of uncontrolled seizures (may be on anticonvulsants, provided seizures are under "reasonable" control and that the patient and family understand the risk of altered seizure control and potential interference with maintaining therapeutic levels of anticonvulsants)
* Hypothyroidism
* Symptoms of affective and mood disorders
* Previously diagnosed with ADHD prior to the onset of neurological complications (e.g., stroke or silent infarct) as documented in the medical record or caregiver report.
* Mental retardation (FSIQ < 70 on WASI)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Conners Parent and teacher Rating Scale | 1 week

SECONDARY OUTCOMES:
Childrens Verbal Learning Test | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T Brown, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina